CLINICAL TRIAL: NCT01096563
Title: A Phase I, Single Centre, Double-blind, Randomised, Placebo-controlled, Parallel-group Study to Assess the Safety, Tolerability and Pharmacokinetics of Inhaled AZD9164 After Administration of Single and Multiple Ascending Doses for 13 Days in Healthy Male and Female Japanese Subjects
Brief Title: A Single and Multiple Ascending Dose Study With AZD9164 Given for 13 Days in Healthy Male and Female Japanese Subjects
Acronym: JSMAD
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor has taken the decision to terminate further development of the compound
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: D1882C00004; 2009-015560-34 (EudraCT Number)
Record Dates: First submitted 2010-03-25; First posted 2010-03-31 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Healthy
Keywords: Phase I; Japanese healthy volunteer; AZD9164
MeSH Terms: interventions — AZD9164

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): AZD9164
  Interventions: Drug: AZD9164
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD9164 — Dry powder for inhalation via Turbuhaler, JSMAD. A single dose of AZD9164 on Day 1 and repeated dosing on Day 4 to day 15 (JSMAD).
  The starting dose will be 400 μg delivered dose and subsequent doses are planned to be 1000 μg and 2800 μg delivered dose.
  Arms: 1
Drug: Placebo — Dry powder for inhalation via Turbuhaler, JSMAD.
  Arms: 2

SUMMARY:
This is a single centre, Double blinded, Randomised, Placebo-controlled, Parallel group study to access the safety, tolerability, and pharmacokinetics of Inhaled AZD9164 after administration of single and Multiple Ascending doses in Japanese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese subjects with suitable veins for cannulation or repeated venipuncture
* Have a body mass index (BMI) between 18 and 27 kg/m2 and a body weight between 50 and 85 kg
* Male subjects should be willing to use barrier contraception ie, condoms with spermicide, from the first day of dosing until 3 months after the last dose of investigational product

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
* History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs
* Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of investigational product

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Safety measurements (ECG's, Telemetry, Pulse, Blood Pressure, Safety Laboratory and Adverse Events) | Safety will be monitored continously and safety assessments will be made on several occasions throughout the whole study

SECONDARY OUTCOMES:
To investigate the pharmacokinetics (PK) of AZD9164 following inhaled administration of single and multiple ascending doses, by assessment of the dose proportionality, the degree of accumulation and the time linearity | PK sampling during the residential period and intense PK sampling on day 1 and day 15 (up to 72 and 120 hours respectively)
To investigate pharmacodynamic (PD) effects of inhaled single and multiple ascending doses of AZD9164, by assessment of lung function | Spirometry during the residential stay on days 1, 4, 6, 7, 8, 9, 10, 11, 12, 13, 14, and 15

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Lorch, MD MFPM FRCA, Principal Investigator — Richmond Pharmacology Limited; Carin Jorup, Study Director — AstraZeneca
Locations (1):
- Research Site, Croydon, United Kingdom

REFERENCES:
- [Derived] Jorup C, Bengtsson T, Strandgarden K, Sjobring U. Transient paradoxical bronchospasm associated with inhalation of the LAMA AZD9164: analysis of two Phase I, randomised, double-blind, placebo-controlled studies. BMC Pulm Med. 2014 Mar 27;14:52. doi: 10.1186/1471-2466-14-52. PMID 24669829